CLINICAL TRIAL: NCT04059978
Title: Pain Response to Cannabidiol in Opioid-induced Hyperalgesia, Acute Nociceptive Pain and Allodynia By Using a Model Mimicking Acute Pain in Healthy Adults
Acronym: CANAB II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2019-01217; qu18Ruppen3
Record Dates: First submitted 2019-08-12; First posted 2019-08-16 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Acute Nociceptive Pain; Hyperalgesia; Allodynia; Opioid-induced Hyperalgesia
Keywords: Cannabidiol; Remifentanil
MeSH Terms: conditions — Hyperalgesia | interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBD + Remifentanil (Active Comparator): CBD 1600 mg p.o. + Remifentanil 0.1 µg/kg/min i.v. for 30 min
  Interventions: Drug: CBD; Drug: Remifentanil
- Placebo + Remifentanil (Placebo Comparator): Placebo p.o + Remifentanil 0.1 µg/kg/min i.v. for 30 min
  Interventions: Drug: Placebo; Drug: Remifentanil

INTERVENTIONS:
Drug: CBD — 1600mg cannabidiol, single oral dose (8 ml oily solution)
  Arms: CBD + Remifentanil
Drug: Placebo — Placebo p.o, single oral dose (8 ml oily solution)
  Arms: Placebo + Remifentanil
Drug: Remifentanil — Remifentanil 0.1 µg/kg/min i.v. for 30 min

SUMMARY:
Prospective, randomized, placebo-controlled, double-blinded, crossover study to investigate the effect of cannabidiol (CBD) on remifentanil-induced hyperalgesia in healthy volunteers in a well-established acute pain model. Participants are randomized according to the order of the two treatments (CBD + Remifentanil or Placebo + Remifentanil).

DETAILED DESCRIPTION:
Opioid-induced hyperalgesia (OIH) is a clinically often neglected, but well described phenomenon. OIH could also be shown for Remifentanil in an acute pain model. As CBD showed antihyperalgesic potential in the animal model, this brings up the question if CBD might be used to prevent or diminish OIH. Until today there are no studies investigating CBD as an adjunct to remifentanil or other opioids regarding the OIH. This is however of great clinical value because CBD with its possible antihyperalgesic effect on the OIH might be a worthful adjunct for opioid based anaesthesia and analgesia.

Every participant will pass through two interventions with electrically induced pain (Koppert model). CBD will be applied orally at the beginning of the intervention. Pain, allodynia and hyperalgesia will be assessed and recorded every 10 min during the remifentanil infusion and afterwards.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.5 until 25 kg/m2
* Able to give informed consent

Exclusion Criteria:

* Regular consumption of cannabinoids or other drugs / substances
* Regular intake of medications potentially interfering with pain sensation (analgesics, antihistamines, calcium and potassium channel blockers, serotonin / noradrenaline reuptake inhibitors, corticosteroids)
* Neuropathy
* Chronic pain
* Neuromuscular disease
* Psychiatric disease
* Known or suspected kidney or liver disease
* Pregnancy (cf. 8.6 Trial specific preventive measures) / Lactation
* Allergy / hypersensitivity to cannabidiol
* Contraindications for Remifentanil (e.g. hypersensitivity)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-05-26 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Change in hyperalgesia measured by the area under the curve (AUCHyper) | from minute 100 to minute 160 after termination of remifentanil infusion
  Change in hyperalgesia measured by the area under the curve (AUCHyper)

SECONDARY OUTCOMES:
Change in pain response (NRS) measured by the area under the curve (AUCNRS) | from minute 70 to minute 90 during remifentanil infusion
  Change in pain response (NRS) measured by the area under the curve (AUCNRS)
Change in hyperalgesia measured by the area under the curve (AUCHyper) | from minute 70 to minute 90 during remifentanil infusion
  Change in hyperalgesia measured by the area under the curve (AUCHyper)
Change in allodynia measured by the area under the curve (AUCAllo) | from minute 70 to minute 90 during remifentanil infusion
  Change in allodynia measured by the area under the curve (AUCAllo)
Change in pain response (NRS) measured by the area under the curve (AUCNRS) | from minute 100 to minute 160 after termination of remifentanil infusion
  Change in pain response (NRS) measured by the area under the curve (AUCNRS)
Change in allodynia measured by the area under the curve (AUCAllo) | from minute 100 to minute 160 after termination of remifentanil infusion
  Change in allodynia measured by the area under the curve (AUCAllo)

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Schneider, MD, Principal Investigator — Department of Anaesthesiology, University Hospital of Basel
Locations (1):
- Department of Anaesthesiology, University Hospital of Basel (USB), Basel, Switzerland

REFERENCES:
- [Derived] Dieterle M, Zurbriggen L, Mauermann E, Mercer-Chalmers-Bender K, Frei P, Ruppen W, Schneider T. Pain response to cannabidiol in opioid-induced hyperalgesia, acute nociceptive pain, and allodynia using a model mimicking acute pain in healthy adults in a randomized trial (CANAB II). Pain. 2022 Oct 1;163(10):1919-1928. doi: 10.1097/j.pain.0000000000002591. Epub 2022 Jan 24. PMID 35239547